CLINICAL TRIAL: NCT03453320
Title: Infusion Rate and Volume Kinetics for Hyperoncotic Albumine in Healthy Subjects
Acronym: (RAV)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Joachim Zdolsek, MD, PhD, Assoc prof, consultant, University Hospital, Linkoeping
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RAV
Record Dates: First submitted 2018-02-24; First posted 2018-03-05 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Edema Secondary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rapid - Slow (Experimental): Two infusions of 3 ml/kg bodyweight of hyperoncotic albumin 20%, with an interval of 3 to 20 weeks between.
  First time rapid (30 minutes), second time slow (120 minutes). Albumin solution
  Interventions: Drug: Albumin solution
- Slow - Rapid (Experimental): Two infusions of 3 ml/kg bodyweight of hyperoncotic albumin 20%, with an interval of 3 to 20 weeks between.
  First time rapid (120 minutes), second time slow (30 minutes). Albumin solution
  Interventions: Drug: Albumin solution

INTERVENTIONS:
Drug: Albumin solution — Infusion rate and effects

SUMMARY:
Treatment with colloidal solutions has during long time been a cornerstone within intensive care. Lately there has been a shift from synthetic colloids to natural albumine.

One of these solutions is the hyperoncotic "Albumin 20%". There are however still several aspects of the physiological effects of hyperoncotic albumin, that are not known.

In this study the main object is to study with what rate hyperoncotic albumin should be administered. Rapidly 30 minutes or slower 120 minutes.

DETAILED DESCRIPTION:
Difference in volume expansion as well as fluid recruitment from the tissues depending on infusion rate is of interest.

Plasma volume expansion is measured using hemoglobin as a marker and fluid recruitment of tissue fluid is measured as a combination of plasma volume expansion and urinary output.

Healthy individuals are asked to refrain from eating and drinking the night before the study. Two hours before study start, the subjects may take a sandwich and a glas to drink.

After 15 minutes of rest baseline blood samples are taken. Subjects are randomised to receive two rates of albumin solution (Albumin 20%) 3 ml/kg bodyweight at two separate occasions. Once with an infusion time of 30 minutes, once with an infusion time of 120 minutes. Between the two infusions there will be an interval of 3 to 20 weeks. Randomization is performed to chose which rate the subjects start with. 6 in each Group (total 12).

During each occasion15 blood samples are collected, during a 6 hour period. Hemoglobin, plasma Sodium, colloid osmotic pressure and albumin are analysed. The total volume of blood collected will be 170 ml at each occasion when an albumin infusion is given.

Urinary output is measured and Urinary Sodium content is measured. Liberal fluid intake is recommended the same day and the next.

ELIGIBILITY:
Inclusion Criteria:

- Healthy, without allergies and with the age 18 years or above

Exclusion Criteria:

* Heart failure
* Signs of kidney injury/failure
* Severe allergies
* Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-02-24 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Plasma volume | 6 hours
  Albumin infusion expands the plasma volume and dilutes hemoglobin. The dilution of hemoglobin can be measured and is used to calculate the degree of plasma expansion.

SECONDARY OUTCOMES:
Colloid osmotic pressure | 6 hours
  Infusion of hyperoncotic albumin increases the colloid osmotic pressure of plasma. Fluid recruitment from the tissues however diminishes the increase of the colloid osmotic pressure. This effect is measured.
Fluid recruitment from tissues | 6 hours
  The recruitment of fluid from the tissues due to the increase of colloid osmotic pressure is measured. The total recruitment of fluid from the tissues is the sum of the plasma volume dilution and urinary excretion.

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Zdolsek, MD, PhD,Assoc prof, Principal Investigator — University Hospital, Linkoeping
Locations (1):
- Intensive Care Unit, University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Undecided